CLINICAL TRIAL: NCT06943495
Title: PROstate-specific Membrane Antigen DosImetry- Guided endoradiotherapY: A Randomized- Controlled, Single-blind, Pilot Study of Personalized vs. Fixed-activity 177Lu-PSMA-617 Radiopharmaceutical Therapy (PRODIGY-2)
Brief Title: Personalized vs. Fixed-Activity 177Lu-PSMA-617 Radiopharmaceutical Therapy (PRODIGY-2)
Acronym: PRODIGY-2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jean-Mathieu Beauregard (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); Novartis (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Jean-Mathieu Beauregard, Nuclear Medicine Physician, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-7829
Record Dates: First submitted 2025-03-25; First posted 2025-04-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Pluvicto

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Personalized activity (Experimental)
  Interventions: Drug: 177Lu-PSMA-617
- Fixed activity (Active Comparator)
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — 6 cycles of personalized activity (1st cycle based on BSA and eGFR; cycles 2-6 based on renal dosimetry), maximum 22.2 GBq, every 6 weeks
  Arms: Personalized activity
Drug: 177Lu-PSMA-617 — 6 cycles of 7.4 GBq every 6 weeks
  Arms: Fixed activity

SUMMARY:
The goal of this clinical trial is to assess if a personalized regime of 177Lu-PSMA-617 (Lutetium Lu 177 vipivotide tetraxetan, also known as Pluvicto) is feasible and safe in a population of patients with metastatic castrate-resistant prostate cancer (mCRPC). The main questions it aims to answer are:

1. Can the administered activity (cumulative or per-cycle) be increased in a majority of participants?
2. What is the incidence of some specific adverse reactions during the treatment?

Researchers will compare participants receiving a personalized regime to participants receiving the standard fixed-activity regime of 177Lu-PSMA-617 to see if the activity can be safely increased through personalization based on renal dosimetry (i.e. the measure of how much radiation is actually delivered to the kidney).

Participants will receive up to 6 treatments of 177Lu-PSMA-617 every 6 weeks and be regularly evaluated with imaging and laboratory tests, as well as with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥18 years with metastatic adenocarcinoma of the prostate, defined by documented histopathology of prostate adenocarcinoma;
2. Castration-resistant prostate cancer, as defined as disease progressing despite castration by orchiectomy or ongoing androgen deprivation therapy;
3. Progressive mCRPC with rising PSA level, defined by PCWG3 criteria (sequence of two rising values above a baseline at a minimum of 1-week intervals, with serum testosterone level ≤ 1.7 nmol/dL);
4. PSA ≥2 ng/mL ;
5. Prior treatment with at least one ARPI;
6. PSMA-expressing cancer, with significant PSMA expression defined as SUVpeak in at least one lesion that is superior to SUVmean of the liver on PSMA-PET (68Ga-PSMA-11 or 18F-DCFPyL), within 45 days prior to randomization;
7. ECOG Performance status 0 to 2;
8. Calculated eGFR (by CKD-EPI formula) ≥ 45 mL/min/1.73m^2;
9. Albumin ≥ 25 g/L;
10. Platelets ≥ 100x10^9/L;
11. Neutrophils ≥ 1.5x10^9/L;
12. Hemoglobin ≥ 90 g/L without transfusion in the past 4 weeks;
13. Signed, written informed consent

Exclusion Criteria:

1. PSMA-PET "superscan" (i.e. extensive/diffuse PSMA-positive bone involvement);
2. Site(s) of disease that are FDG-positive, defined as SUVpeak in at least one lesion that is superior to twice (2x) SUVmean of the liver, and PSMA-negative (as above), within 45 days prior to randomization;
3. Prior treatment with more than two lines of chemotherapy for mHSPC and/or mCRPC (adjuvant and neoadjuvant chemotherapy does not count) towards the maximum of two regimens);
4. Prior radiopharmaceutical therapy;
5. Known CNS metastasis unless they are deemed to be non-progressive, asymptomatic and off corticosteroid therapy for at least four weeks, as per investigator's assessment;
6. Active malignancy other than prostate cancer;
7. Patients who are sexually active and not willing/able to use medically acceptable forms of barrier contraception;
8. Any other condition, diagnosis or finding that may in the investigator's opinion interfere with trial conduct;
9. Known hypersensitivity to 177Lu-PSMA-617 or to any ingredient in the formulation, including any non-medicinal ingredient, or component of the container.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Administered activity of 177Lu-PSMA-617 | From first administration to the end of treatment (each cycle is 6 weeks, up to 6 cycles)
  In GBq, cumulative and average per cycle.
Number of participants with subacute adverse events of special interest (AESIs) | From first administration to the end of treatment (each cycle is 6 weeks, up to 6 cycles)
  Subacute AESIs are:
  * treatment-related grade 3-4 thrombopenia persisting more than 12 weeks
  * treatment-related grade 3-4 neutropenia persisting more than 12 weeks
  * treatment-related creatinine elevation to >2x baseline and >ULN (upper limit of normal) persisting more than 12 weeks
  * treatment-related grade 4 febrile neutropenia
  * treatment-related grade 4 non-hematological toxicity

SECONDARY OUTCOMES:
Best biochemical response | From first administration until 52 weeks or the start of another anti-cancer treatment or death, whichever is earliest
  Maximum percent decrease of serum prostate-specific antigen (PSA) after first administration.
PSA progression-free survival (PSA-PFS) | From date of first administration until the date of PSA progression or of the start of another anti-cancer treatment or of death, whichever came first, assessed over a minimum of 60 months
  Time from first administration to an increase in PSA greater than 25%, and greater than 2 ng/ml, above nadir, confirmed at least 3 weeks later.
Best radiological response rates | From first administration to the end of treatment (each cycle is 6 weeks, up to 6 cycles)
  Percentage of participants achieving each RECIST 1.1 response category as their best response: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), overall response (i.e., CR or PR; a.k.a. overall response rate, ORR), disease control (i.e CR, PR or SD; a.k.a. disease control rate, DCR).
Radiological progression-free survival (rPFS) | From date of first administration until the date of radiological progression or of the start of another anti-cancer treatment or of death, whichever came first, assessed over a minimum of 60 months
  Time from first administration to the date of radiographic disease progression based on RECIST 1.1/PCWG3.
Investigator-assessed overall PFS | From date of first administration until the date of investigator-assessed progression or of the start of another anti-cancer treatment or of death, whichever came first, assessed over a minimum of 60 months
  Time from first administration to the earliest of clinical (worsening of a patient's clinical status attributed to disease progression), biochemical or radiological progression considering all data (scheduled and unscheduled) available to the investigator.
Time to first symptomatic skeletal event (SSE) | From date of first administration until the date of first SSE or of the start of another anti-cancer treatment or of death, whichever came first, assessed over a minimum of 60 months
  Time to first Symptomatic Skeletal Event (SSE) is defined as the time from first administration to the date of the SSE. The SSE date is the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever occurred first.
Overall survival (OS) | From date of first administration until the date of death, assessed over a minimum of 60 months
  Overall Survival (OS) is defined as the time from the date of the first administration to the date of death due to any cause.
Metabolic response on FDG-PET/CT | At baseline and at 12 weeks
  Metabolic response is defined as complete metabolic response (CMR, disappearance of all lesions on FDG PET), partial metabolic response (PMR, decrease of uptake by ≥30%), stable metabolic disease (SMD, variation of FDG uptake by <30%), progressive metabolic disease (PMD, increase of FDG uptake by ≥30%)
Molecular response on PSMA-PET/CT | At baseline and at the end of treatment (each cycle is 6 weeks, up to 6 consecutive cycles)
  Molecular response is defined as the variation of molecular tumor volume (MTV) on PSMA-PET/CT
Best molecular response on quantitative 177Lu SPECT/CT during treatment | From first cycle's Day 3 until the last cycle's Day 3 (each cycle is 6 weeks, up to 6 consecutive cycles)
  Best molecular response is defined as the maximum percent decrease of molecular tumor volume (MTV) at any time after post-treatment quantitative 177Lu SPECT/CT performed on the first cycle's Day 3, up to the post-treatment quantitative 177Lu SPECT/CT performed on the last cycle's Day 3
Number of participants with any adverse events (AEs) | From first administration to the end of treatment (each cycle is 6 weeks, up to 6 cycles)
  All adverse events that occur from the first administration of 177Lu-PSMA-617 until 6 weeks after the last administration of 177Lu-PSMA-617 or prior to the initiation of subsequent anticancer treatment.
Number of participants with laboratory adverse events (AEs) | From date of first administration until the date of investigator-assessed progression or of the start of another anti-cancer treatment or of death, whichever came first, assessed over a minimum of 60 months
  Adverse events seen on laboratory (hematology, biochemistry) that occur from the first administration of 177Lu-PSMA-617 until progression or until the initiation of subsequent anticancer treatment if earlier.
Number of participants with delayed adverse events of special interest (AESIs) | From date of first administration until the date of death, assessed over a minimum of 60 months
  Delayed AESIs (renal impairment and secondary hematological malignancies) that occur from the first administration of 177Lu-PSMA-617 until death (or study termination)
Variation of score on EuroQol-5 Dimension-5 Level (EQ-5D-5L) questionnaire at baseline | At baseline, at 18 weeks, and at the end of treatment (each cycle is 6 weeks, up to 6 consecutive cycles)
Variation of score on Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire at baseline | At baseline, at 18 weeks, and at the end of treatment (each cycle is 6 weeks, up to 6 consecutive cycles)
Variation of score on Brief Pain Inventory (BPI-SF) questionnaire at baseline | At baseline, at 18 weeks, and at the end of treatment (each cycle is 6 weeks, up to 6 consecutive cycles)
Variation of score on Multidisciplinary Salivary Gland Society (MSGS) questionnaire at baseline | At baseline, at 18 weeks, and at the end of treatment (each cycle is 6 weeks, up to 6 consecutive cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Mathieu Beauregard, MD, Principal Investigator — CHU de Québec-Université Laval
Locations (1):
- CHU de Québec-Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There is an intent to create an imaging and data bank from this study.